CLINICAL TRIAL: NCT01211886
Title: Utility of BNP in Patients With Type IV Cardio-renal Syndrome Admitted to the ICU: a Prospective Observational Study
Brief Title: Utility of Brain Natriuretic Peptide (BNP) in Patients With Type IV Cardio-renal Syndrome Admitted to the Intensive Care Unit (ICU)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: f2000tj1
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Kidney Disease; Acute Heart Failure
Keywords: Brain natriuretic peptide; Cardio-renal syndrome
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardio-Renal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum sample for BNP level
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Admission BNP was a useful marker for diagnosing and predicting type IV cardio-renal syndrome type IV in patients with chronic kidney disease admitted to the ICU for acute heart failure in a retrospective study. Therefore, we aim to prospectively investigate the utility of serum BNP in evaluating the treatment adequacy and predicting future cardiac events in patients with type IV CRS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged > 18 years, Patients with chronic kidney disease (Serum Cr > 2.0, Documented medical history of chronic kidney disease

Exclusion Criteria:

* Cardiopulmonary resuscitation, Do-not-resuscitate state, Acute kidney injury, ICU stay < 1 day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease admitted to the ICU for acute heart failure (i.e., type IV cardio-renal syndrome)
Sampling Method: Non-Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-08 (Estimated)